CLINICAL TRIAL: NCT05404893
Title: Fecal Calprotectin Levels in Patients With Fibromyalgia: A Cross-sectional Study
Brief Title: Fecal Calprotectin Levels in Patients With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Principal investigator, Ege University
Other Study IDs: Ege 20-10T/47
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Abdominal Pain
Keywords: fecal calprotectin; fibromyalgia; irritable bowel syndrome; abdominal pain
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fibromyalgia without gastrointestinal symptoms: Patients diagnosed as having Fibromyalgia according to american college of rheumatology 2016 classification criteria, with no abdominal pain, constipation, diarrhea, tenesmus, abdominal cramps
  Interventions: Diagnostic Test: Fecal calprotectin measurement
- Fibromyalgia with gastrointestinal symptoms: Patients diagnosed as having Fibromyalgia according to american college of rheumatology 2016 classification criteria, with abdominal pain and constipation and/or diarrhea and/or tenesmus and/or abdominal cramps
  Interventions: Diagnostic Test: Fecal calprotectin measurement
- Healthy controls: Healthy controls, no gastrointestinal symptoms
  Interventions: Diagnostic Test: Fecal calprotectin measurement

INTERVENTIONS:
Diagnostic Test: Fecal calprotectin measurement — Stool samples will be collected and fecal calprotectin levels will be measured using an enzymatic immunoassay kit.

SUMMARY:
This study was designed to evaluate fecal calprotectin levels in patients with fibromyalgia syndrome. Fecal calprotectin levels from fibromyalgia patients with and without gastrointestinal symptoms as well as healthy controls will be measured and compared.

DETAILED DESCRIPTION:
Fecal calprotectin (FC) is a calcium and zinc binding protein that is present in neutrophil granulocytes and is detected in the stool samples from subjects with inflammatory bowel disease and similar organic gastrointestinal pathologies. Fibromyalgia is often accompanied by irritable bowel syndrome, which is a non-inflammatory, functional disorder of the gastrointestinal tract. Due to the chronic nature of the disease, fibromyalgia patients' new symptoms related to underlying gastrointestinal organic disease may be overlooked. In this study we aimed to assess the FC levels in fibromyalgia patients and healthy controls in order to detect a possible difference in FC levels between patients with and without gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Groups 1 and 2: patients diagnosed as having Fibromyalgia syndrome according to American College of Rheumatology 2016 classification criteria (8). Group 3 will consist of healthy controls
* Older than 18 years of age

Exclusion Criteria:

* Presence of gastrointestinal symptoms starting after the age of 50.
* Presence of inflammatory rheumatological disorder
* Presence of organic gastrointestinal disorder
* History of fever, infective gastroenteritis, endoscopy or colonoscopy in the previous month
* Family history of inflammatory bowel disease
* Patients with alarm symptoms that required further investigation such as weight loss, nocturnal diarrhea, rectal bleeding
* Illiteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects diagnosed as having FMS according to American College of Rheumatology 2016 classification criteria (1). Group 3 will consist of healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Fecal calprotectin levels | 1 day
  Fecal calprotectin levels higher than 50 microgram/grams of feces will be considered positive

SECONDARY OUTCOMES:
Correlation of fecal calprotectin levels with fibromyalgia disease parameters | 1 day
  Fecal calprotectin levels will be assessed for correlation with symptom severity scale and widespread pain index scores of american college of rheumatology 2016 classification criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ece Cinar, MD, Principal Investigator — Ege university school of medicine; Burcu Turkoglu Aytar, MD, Study Chair — Kirsehir Ahievran University School of Medicine; Simin Hepguler, Prof., Study Chair — Ege university school of medicine; Burcu Barutcuoglu, Ass.Prof., Study Chair — Ege university school of medicine
Locations (1):
- Ege University School of Medicine, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Ayling RM, Kok K. Fecal Calprotectin. Adv Clin Chem. 2018;87:161-190. doi: 10.1016/bs.acc.2018.07.005. Epub 2018 Oct 1. PMID 30342711